CLINICAL TRIAL: NCT01677416
Title: Joint Ultrasound Evaluation of Asymptomatic Feet in Patients With Rheumatoid Arthritis: A Controlled Study
Brief Title: Joint Ultrasound Evaluation of Asymptomatic Rheumatic Feet
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Anamaria Jones, Principal Investigator, Federal University of São Paulo
Other Study IDs: UNIFESP/2011
Record Dates: First submitted 2012-08-27; First posted 2012-09-03 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Ultrasonography; Synovitis; Foot joints
MeSH Terms: conditions — Arthritis, Rheumatoid; Synovitis

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis Group: RA with at least one year since diagnosis, asymptomatic feet, and age between 18 and 65 years
- Control group: Absence of known osteoarticular disease

SUMMARY:
Objectives: The aims of the present study were to compare ultrasound on asymptomatic feet of patients with rheumatoid arthritis (RA) and normal controls, determine the association between ultrasound and global disease activity, function and goniometric measures in patients with RA and determine the correlation between ultrasound and radiography in the detection of bone erosion.

Methods: The foot joints (talocrural, talocalcaneal, talonavicular, naviculocuneiform, calcaneocuboid, 5th tarsometatarsal and 1st to 5th metatarsophalangeal [MTP] joints) of 50 healthy subjects and 50 patients with RA (all with asymptomatic feet) were evaluated bilaterally regarding quantitative/semi-quantitative synovitis, semi-quantitative Power Doppler (PD) signals and erosion using ultrasound. Statistical significance was set to 5%.

ELIGIBILITY:
Inclusion Criteria:

Rheumatoid Arthritis Group:

* RA with at least one year since diagnosis
* Asymptomatic feet
* Age between 18 and 65 years Control group
* absence of known osteoarticular disease

Exclusion Criteria for both groups:

* Peripheral venous insufficiency with retrograde venous flow and/or ochre dermatitis
* Previous surgical intervention and/or fracture in feet/ankles
* Intra-articular corticosteroid injection in previous three months in any of the joints evaluated
* Foot neuropathy
* Pain and swelling in feet or ankles

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Rheumatoid Arthritis
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Presence of synovial effusion and/or synovial hypertrophy | Baseline
  Ultrasound evaluation - quantitative measurement considered the distance between the joint capsule and subchondral bone of the joints studied (talocrural, talocalcaneal (medial, lateral and posterior windows); dorsal face of calcaneocuboid, talonavicular, medial naviculocuneiform, 5th tarsometatarsal and metatarsophalangeal (MTP) (dorsal and volar faces of 1st to 5th MTP joints and lateral face of 1st and 5th MTP joints). A modified score was used for the semi-quantitative measurement, ranging from 0 to 3: 0-no synovial thickening; 1-minimal synovial thickening in joint recess; 2-synovial thickening in entire joint recess causing bulging of joint capsule; and 3-synovial thickening in joint recess with bulging of joint capsule and extending to at least one bone diaphysis. "Presence of synovitis" was defined as synovial hypertrophy of at least Grade 1 in the semi-quantitative analysis (gray scale - ultrasound)
Presence of bone erosion | Baseline
  defined based on the preliminary OMERACT criteria: intra-articular discontinuity of the bone surface observed on two perpendicular planes. A previously established semi-quantitative score (0-3) was employed: 0-uniform bone surface; 1-irregular bone surface; 2-bone surface defect on two planes; 3-bone defect causing extensive bone destruction. The "presence of erosion" was defined as the presence of at least Grade 2 erosion.

SECONDARY OUTCOMES:
Radiographic evaluation | Baseline
  A blinded radiologist analysed the presence of erosion in each joint studied. For such, ankle (AP and profile) and foot (AP and profile with load) radiographs were taken.
Intraobserver and interobserver agreement | Baseline
  The patients with RA were submitted to clinical and ultrasound evaluations of the feet and ankles on the same day. The ultrasound measurements intraobserver/interobserver agreement was performed on the talocrural, talonavicular and 5th MTP joints, using 20% of the sample. For this, the ultrasound exams were performed by another rheumatologist.
Presence of synovial blood flow | Baseline
  The presence of Power Doppler (PD) signals was evaluated in the bone margins, joint spaces, and peri-articular tissues (frequency of 8 MHz and pulse repetition rate of 750 MHz). A semi-quantitative score (0-3) was employed[14]: 0-no signal; 1-minimal signal, presence of simple vessels; 2-moderate signal, presence of confluent vessels with signal in less than 50% of the area evaluated; 3-intense signal (more than 50% of area evaluated). "Active synovitis" or "presence of PD signal" was defined as the presence of intra-articular synovitis with a positive PD signal (at least Grade 1).

CONTACTS AND LOCATIONS:
Overall Officials: Rita Furtado, MD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Universidade Federal de Sao Paulo, São Paulo, SP - Sao Paulo, Brazil